

### CONSENT TO PARTICIPATE IN A CLINICAL RESEARCH STUDY

**STUDY TITLE:** Omega Heroes: Fatty Acid Supplements and Inflammation in Children with

Autsim Spectrum Disorder

PRINCIPAL INVESTIGATOR: Dr. Sarah Keim

**CONTACT TELEPHONE NUMBER:** 614-355-2849; 1-800-792-8401, extension 52849

STUDY SPONSOR: National Institutes of Health, National Center for Complementary and Integrative

Health

| SUBJECT'S NAME: | DATE OF BIRTH: |
|-----------------|----------------|
|-----------------|----------------|

NOTE: The words "you" and "your" are used in this consent form. These words refer to the study volunteer whether a child or an adult.

## **Key Information About This Study**

The following is a short summary of this study to help you decide whether or not to participate. More detailed information follows later in this form.

The purpose of this study is to find out if a fatty acid nutritional supplement oil is an effective treatment for autism spectrum disorder symptoms.

### Study participation:

You will be asked to give your child a fatty acid nutritional supplement oil or placebo oil every day (in the morning and evening) for 3 months.

Your child will have blood drawn 3 times during participation.

You will be asked to complete some questionnaires.

Your child will be asked to do autism assessments.

You will complete a study diary to show if your child took the oil each day.

### Study visits:

There will be 3 visits over 3 months at the main campus of Nationwide Children's Hospital.

First visit: 3 hours, second visit: 1 hour, third visit: 3 hours

We will call you about five times within the 3 months of participation. One call will last longer (20-25 minutes) than the others.

See a more detailed discussion later in this form.

The main risks of the study are bleeding and bruising at the site where the blood is drawn, allergic reaction to nutritional supplement oil or placebo oil, and mild diarrhea, gas or other intestinal related symptoms associated with nutritional supplement oil or placebo oil.

You and your child may not benefit from being in this study. We hope that the information learned will help others in the future who have an autism spectrum disorder diagnosis.

If you are interested in learning more about this study, please continue reading below.



## 1) INTRODUCTION

This is a research study that is interested in learning about how a nutritional supplement oil may help children with Autism Spectrum Disorder (ASD). Dr. Sarah Keim and Dr. Lynette Rogers are working on this study with doctors from the Developmental and Behavioral Pediatrics Department at Nationwide Children's Hospital. We invite you to participate in this research study because your child was recently diagnosed with ASD.

Using this form as a guide, we will explain the study to you. If you have any questions about the study, please ask. By signing this form, you agree to be in this study. If you do not want to be in this study, all regular and standard medical care will still be available to you here at Nationwide Children's Hospital. Participation is voluntary. You can leave this study at any time.

You will be given a signed and dated copy of the consent form.

# 2) WHERE WILL THE STUDY BE DONE AND HOW MANY SUBJECTS WILL TAKE PART?

This study will be done at Nationwide Children's Hospital and we hope to enroll 98 participants.

## 3) WHAT WILL HAPPEN DURING THE STUDY AND HOW LONG WILL IT LAST?

This study will last for 90 days, about 3 months.

During the study, we ask that you give your child a nutritional supplement oil or placebo oil every day, twice a day, during the study. We also ask that you come to Nationwide Children's Hospital 3 times. Visit 1 is today. Visit 2 will be 45 days later and visit 3 will be 45 days after that. If you have a visit scheduled already in any of the Nationwide Children's Hospital clinics, we will try to make the study visit the same day to make it convenient. The first and last study visits would last about 3 hours. The second study visit will last about 1 hour.

## What we ask you to do:

- During the study visits, we will ask you to answer questions about your child's diet and your family. You have the option of skipping any question you do not want to answer. We will ask you to provide us with updated contact information. We will not share this information with anyone outside the research team and we will only contact you about the study.
- During the first and last in-person visits, trained research staff will:
  - 1) measure your child's height and weight
  - complete some development and behavior assessments with you and your child
  - 3) complete a questionnaire about your child's gastrointestinal history (stomach problems)
- During each in-person visit, a 3mL (about half a teaspoon) blood sample will be drawn from a
  vein in your child's arm by an experienced and trained Nationwide Children's Hospital
  employee. The blood drawn during each visit will be used to see how much of the oil your
  child is taking and how the body is responding to the oil.



- At the first study visit, you will be given bottles of an oil to take home with you. We will ask you
  to give your child the oil each day. We will provide a study diary and instructions for you to
  record that your child took the oil.
- We will check in with you about 5 times to see how the study is going for you. One of these
  phone calls will request a more detailed update than the others. We will call this phone call our
  "e-visit." We will provide you with our phone number and e-mail address for you to contact us
  with any concerns or questions. During the follow up calls, study staff will request photos of
  complete study diary pages on occasion. These photos can be texted or emailed on the day of
  the follow up call.

To check to see if the fatty acids help children with ASD we need different groups of families. To determine which group each family is in, this study is randomized. Randomized means that each family will be picked by chance, like tossing a coin or drawing straws, to receive either the fatty acid supplement oil or placebo oil. Each subject has a 50/50 chance of receiving the fatty acid supplement oil and a 50/50 chance of receiving the placebo oil. By randomizing families into one of the groups, we can check in a fair way to see if the nutritional supplement helps children with ASD.

One group will receive the nutritional supplement which is a liquid that contains oil from fish and oil from a plant called borage. The fatty acids in this liquid are naturally occurring and are found in breast milk and foods like chicken, fish, and cooking oils. The other group will receive a placebo liquid which contains canola oil, a common cooking oil. The nutritional supplement and placebo contain a small amount of lemon to make them taste good. There are no known benefits of the placebo oil. Both the nutritional supplement oil and placebo oil look, smell, and taste the same. You will not know whether you are taking the study medicine or the placebo.

This study is blinded. Blinded means you and all the staff involved in the study will not know who is receiving the nutritional supplement oil or the placebo oil. However, in the case of a medical emergency, there is a way for the study staff to quickly find out which one a child is receiving.

## 4) WHAT ARE THE RISKS OF BEING IN THIS STUDY?

We believe that there is very little chance that bad things will happen as a result of being in this study. It is possible that you could feel upset when answering questions about your child's diagnosis or medical treatment, but it may be more likely that you find the questions or feedback process a little boring. If you do find any of the questions upsetting or don't want to answer a question, you don't have to, and the study team will be available to discuss this with you further.

Although the nutritional supplement oil and placebo oil used in this study are available to buy over-the-counter in local stores, all nutritional supplements or oils may cause some side effects or other reactions. The side effects and discomforts most commonly associated with the medicine and procedures used in this study are listed below. There is no way to give absolute assurance that you will or will not experience any of these or other side effects.

The common side effects may include mild cases of diarrhea, gas or other intestinal related symptoms. Allergic reactions can happen with any nutritional supplement. Symptoms of an allergic reaction can include rash, itching, hives, headache, stomach discomfort, or difficulty breathing.



Because of this, children with a fish, canola, or borage seed allergy are not eligible to participate. Allergic reactions can be severe and possibly life threatening. Severe allergic reactions are a rare possibility.

If any of the symptoms listed above are severe, you must get medical help right away.

If you are worried about anything while in this study, please call the study team at the number on page 1 of this form.

Drawing blood by placing a needle in a vein may cause pain, lightheadedness, fainting, bleeding, bruising, or swelling at the puncture site. Infection is a rare possibility. If needed, numbing cream may be used on the skin to decrease the discomfort. Skin irritation or an allergic reaction is possible from the numbing cream.

Although we will take every precaution, there is a small chance of loss of confidentiality of your study information.

There may be other risks of being in this research study that are not known at this time.

## 5) ARE THERE BENEFITS TO TAKING PART IN THIS STUDY?

Although there may be no benefit to you from being in this study, we hope to learn something that could help other children with ASD and their families in the future.

## 6) WHAT OTHER TREATMENTS OR OPTIONS ARE THERE?

Your participation is this study is voluntary. It is not necessary to participate in this study in order for you to get care for your condition. If you decide not to be in this study, the study team will refer you to your regular doctor for care.

### 7) WHAT ARE THE COSTS AND REIMBURSEMENTS?

It will not cost you anything to be in this study. We will not bill you or your insurance company for the study. For your time and inconvenience, you will be compensated \$85 at the end of each of the 3 inperson study visits. In addition, we will give you \$2 every time you return a study diary (up to \$26 total if all diaries are returned) to thank you for your time and effort. We will pay for your parking in the Children's Hospital Parking Garage during your study visits. We also will give your child a book or toy to take home at the completion of each study visit. If you complete all study visits and the e-visit phone call, you will be compensated an additional \$25 at the end of the final visit.

Additionally, we have a \$125 drawing once per year. You receive entries into the drawing for completing study activities. You can receive up to 15 entries into the drawing. You receive one entry into the drawing for each of the following study activities:

- 1. Return of weekly study diary to study staff.
- 2. Return all of your used and unused bottles of oil.



In regards to your compensation, Nationwide Children's Hospital is now using a service called ClinCard® by the company Greenphire to manage payments for study participation. You will no longer be receiving compensation in cash, check, or by gift card.

You will be issued a ClinCard® debit card specially designed for clinical research. When each study visit is completed, funds will be approved and automatically loaded onto your card. The funds will be available immediately after being loaded, but could take up to 1-2 business days. These funds can be used at your discretion. You will be issued one card for the duration of your participation. If your card is lost or stolen, please call the study coordinator for a replacement card.

Your name, subject number, address, email address, cell phone number and social security number will be collected by Nationwide Children's Hospital in order to issue the debit cards. Debit cards are managed by Greenphire Inc. All information is stored in a secure fashion. Your information will not be shared with any third parties and will be kept completely confidential.

If you receive \$600 or more in a calendar year from participating in research studies, you will be issued a 1099 IRS Form to file with your income taxes.

## 8) WHAT HAPPENS IF BEING IN THIS STUDY CAUSES INJURIES?

We believe that there is very little chance that injuries will happen as a result of being in this study.

If your child is hurt by the nutritional supplement oil or placebo oil or the procedures that are part of this study, you should seek medical treatment for the injuries and call the study team as soon as possible at the number on page 1 of this form. If it is an emergency, call 911 or go to the nearest emergency department.

In most cases, this care will be billed to your health insurance company or whoever usually pays for your health care at the usual charges, but some insurance companies will not pay for care related to a study. If the care is provided at Nationwide Children's Hospital, we make no commitment to pay for the medical care provided to you. No funds have been set aside to compensate you in the event of injury. If no one else pays for your care, you may have to pay for the cost of this care. This does not mean that you give up any of your legal rights to seek compensation for your injuries.

# 9) WHAT WILL HAPPEN IF NEW INFORMATION IS FOUND OUT ABOUT THE DRUG OR TREATMENT?

If new information is found out during this study that might change your mind about participating or might affect your health, the study team will discuss it with you as soon as possible.

## 10) WHAT HAPPENS IF I DO NOT FINISH THIS STUDY?

It is your choice to be in this study. You may decide to stop being in this study at any time. If you decide to stop being in this study, call the study team at the number on page 1 of this form to see if there are any medical issues about stopping. If you stop being in the study, there will be no penalty or loss of benefits to which you are otherwise entitled.



If at any time the Principal Investigator believes that this study is not good for you, the study team will contact you about stopping. If the study instructions are not followed, participation in the study may also be stopped. If unexpected medical problems come up, the Principal Investigator or the Sponsors, National Institutes of Health and National Center for Complementary and Integrative Health, may decide to stop your participation in the study.

## 11) OTHER IMPORTANT INFORMATION

It is important that health care providers know about all medicines that your child is taking. This includes the nutritional supplement oil being tested in this research study. Because of this, we may inform your primary care doctor (if you have one) that your child is participating in this study and document his/her participation in this study in your Nationwide Children's Hospital medical record. This is done so extra care can be taken in prescribing other medicines and looking at any unexplained symptoms that may occur.

| Primary | y Care Physician Contact Info: Name: |
|---------|---------------------------------------|
| | Location (City, State): |
| | Phone Number (including area code): |

Being in more than one research study at the same time may cause injury. Tell us if you are in any other research studies.

If you are an employee of Nationwide Children's Hospital or the Research Institute at Nationwide Children's Hospital, your job or performance appraisal will not be affected in any way if you decline to participate or withdraw your consent to participate in this study.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Website will not include information that can identify you. At most, the Website will include a summary of the results. You can search this Web site at any time.

The final study results will not be shared with you individually. However, at some time, a final study summary will be available on the ClinicalTrials.Gov (http://clinicaltrials.gov) website.

Nationwide Children's Hospital is a teaching hospital and we are committed to doing research. Doing research will enable us to learn and provide the best care for our patients and families. You may be asked to participate in other research studies in the future. You have the right to decide to participate or decline to participate in any future studies. We will not share your contact information with researchers outside Nationwide Children's Hospital.

If study staff observes something that makes us concerned for your welfare or the welfare of your child, we may not be able to keep that information private and will contact the appropriate authorities.



# 12) HOW WILL MY STUDY INFORMATION BE KEPT PRIVATE?

Information collected for this study includes information that can identify you. This is called "protected health information" or PHI. By agreeing to be in this study, you are giving permission to the study team to use or disclose (release) your health information that identifies you for the research study described in this form. Information collected is the property of Nationwide Children's Hospital, its affiliated entities, and/or the sponsor.

**PHI that may be used or disclosed will include:** demographic information such as names, addresses, telephone numbers; medical diagnoses, dates such as admission/discharge and birthdate; and identifying numbers such as medical records number.

# People or Companies authorized to use, disclose, and receive PHI collected or created by this research study:

- The Principal Investigators, Study Doctor, and the study staff
- Representatives of the Office for Human Research Protections, the federal government office that oversees human subject research
- Members of Nationwide Children's Hospital Institutional Review Board (IRB), a committee that reviews all human subjects research for Nationwide Children's Hospital.
- Nationwide Children's Hospital internal auditors
- The Food and Drug Administration (FDA)

Because of the need to give information to these people, absolute confidentiality cannot be guaranteed. Information given to these people may be further disclosed by them and no longer be protected by federal privacy rules.

**Reason(s) why the use or disclosure is being made:** to access medical charts and/or to contact you in the future.

You may decide not to authorize the use and disclosure of your PHI. However, if it is needed for this study, you will not be able to be in this study. If you agree to be in this study and later decide to withdraw your participation, you may withdraw your authorization to use your PHI. This request must be made in writing to the Principal Investigator at:

Sarah Keim, PhD, MA, MS
The Research Institute at Nationwide Children's Hospital
Center for Biobehavioral Health
700 Children's Drive
Columbus, Ohio 43205

If you withdraw your authorization, no new PHI may be collected and the PHI already collected may not be used unless it has already been used or is needed to complete the study analysis and reports.

PHI will only be shared with the groups listed above, but if you have a bad outcome or adverse event from being in this study, the study team or other health care providers may need to look at your entire medical records.



The results from this study may be published but your identity will not be revealed.

A copy of this form and other research related health information may be added to your NCH medical record.

The PHI collected or created under this research study will be used or disclosed as needed until the end of the study. The records of this study will be kept for an indefinite period of time and your authorization to use or disclose your PHI will not expire.

# **Publically Available Scientific Databases**

Some of your specimens and genetic and/or health information might also be placed into one or more external publicly-accessible scientific databases. For example, the National Institutes of Health (an agency of the federal government) maintains a database called "dbGaP." Your name and other information that could directly identify you (such as your address or social security number) will never be placed into these external databases. A researcher who wants to study information from these databases must have an approved study and work with the group overseeing the database to obtain the information. Because it is possible to re-identify de-identified genomic data, even if access to data is controlled and data security standards are met, confidentiality cannot be guaranteed.

## **Certificate of Confidentiality**

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. This means that the researchers cannot release or use information, documents, or samples that may identify you in any action or suit unless you say it is okay. They also cannot provide them as evidence unless you have agreed. This protection includes federal, state, or local civil, criminal, administrative, legislative, or other proceedings. An example would be a court subpoena.

There are some important things that you need to know. The Certificate DOES NOT stop reporting that federal, state or local laws require. Some examples are laws that require reporting of child or elder abuse, some communicable diseases, and threats to harm yourself or others. The Certificate CANNOT BE USED to stop a sponsoring United States federal or state government agency from checking records or evaluating programs. The Certificate DOES NOT stop disclosures required by the federal Food and Drug Administration (FDA). The Certificate also DOES NOT prevent your information from being used for other research if allowed by federal regulations.

Researchers may release information about you when you say it is okay. For example, you may give them permission to release information to insurers, medical providers or any other persons not connected with the research. The Certificate of Confidentiality does not stop you from willingly releasing information about your involvement in this research. It also does not prevent you from having access to your own information.

## 13) USE OF INFORMATION/SAMPLES FOR FUTURE RESEARCH USE

### **Future Research Use of Identifiable Information:**



With your permission, we would like to store your identifiable information (including PHI) for future research purposes, and as part of such future research purposes, your identifiable information may be disclosed to people or entities not listed above, such as researchers not involved with this study, government agencies, research foundations, or pharmaceutical or device companies. This future research may or may not be related to your medical problem. This future research may include sensitive information. Any future research projects will be reviewed and approved by an Institutional Review Board which protects the rights, welfare, and safety of human research subjects. If your identifiable information including PHI is used or disclosed in future research studies, absolute confidentiality cannot be guaranteed. Information shared for future research may be shared further with others and no longer be protected by federal privacy rules.

If you decide at any time that you do not want your PHI stored for future research, you must make this request in writing to the Principal Investigator at:

Sarah Keim, PhD, MA, MS
The Research Institute at Nationwide Children's Hospital
Center for Biobehavioral Health
700 Children's Drive
Columbus. Ohio 43205

Once we receive your written request, we will destroy your PHI. However, if we have already shared your PHI with another individual or entity, we will not be able to destroy any of the PHI that are no longer in our possession.

Nationwide Children's Hospital retains the right to cease storage and destroy the PHI at any time without sending notice to you or obtaining your consent.

You do not have to agree to use of your PHI for future research in order to be in this study, and your decision will not affect the care you receive from the study doctors or Nationwide Children's Hospital.

| I agree to allo | ow my PHI to be | e stored and us | ed for future r | esearch as d | escribed abo | ove: (initial) |
|---|---|---|---|---|---|---|
| YES_ | NO | | | | | |

## **Future Research Use of identifiable Samples:**

Sometimes, a small amount of blood may be leftover from the study and stored for research at a later time, perhaps even years from now.

With your permission, we would like to store unused study samples and information related to such samples (diagnosis, age at diagnosis, etc.) for research that may be performed in the future. Any unused samples will be stored for an indefinite amount of time. Information related to the samples may or may not include personal identifiers, such as your name, address, etc. There could be widespread sharing of these samples and associated information, but an Institutional Review Board, which protects the rights, welfare, and safety of human research subjects, will review and approve each new project.



Use of your samples for future research may help researchers learn more about how to prevent, find, and treat various diseases and conditions, even diseases and conditions that are different from yours. Genetic material (such as DNA and RNA) may be removed from the stored samples and used for genetic testing.

Using your samples for future research will probably not help you. You will not be told the results of any future research. Your doctor will also not be told the results of any future research.

Your samples and information will be used only for research and will not be sold. There is a possibility that future research may lead to development of products that will be sold to the public. If this happens, there is no plan to share any financial gain with you.

The results from this future research may be published but your identity will not be revealed.

If you decide at any time that you do not want your samples or related information stored for future research, you must make this request in writing to the Principal Investigator at:

Sarah Keim, PhD, MA, MS
The Research Institute at Nationwide Children's Hospital
Center for Biobehavioral Health
700 Children's Drive
Columbus, Ohio 43205

Once we receive your written request, we will destroy your samples and related information. However, once your samples and related information have been de-identified, we will not be able to destroy them because we will not be able to link your samples or information back to you. Also, if we have already shared your samples or information with another individual or entity, we will not be able to destroy any of the samples or information that are no longer in our possession.

Nationwide Children's Hospital retains the right to cease storage of the samples or related information at any time and destroy the samples or information without sending notice to you or obtaining your consent.

You do not have to agree to use of your samples or related information for future research in order to be in this study, and your decision will not affect the care you receive from the study doctors or Nationwide Children's Hospital.

| 0 | my samples<br>: (initial your o | information | to be | stored | and | used | for | future | research | n as |
|---|---|---|---|---|---|---|---|---|---|---|
| YES | NO | | | | | | | | | |

## 14) WHOM SHOULD I CALL IF I HAVE QUESTIONS OR PROBLEMS?



If you have questions, concerns, or complaints about anything while on this study or you have been injured by the research, you have 24 hour access to talk to the Principal Investigator or Study Coordinator at 614-355-2849 or 1-800-792-8401, extension 52849.

If you have questions, concerns, or complaints about the research; if you have questions about your rights as a research volunteer; if you cannot reach the Principal Investigator; or if you want to call someone else, call (614) 722-2708, Nationwide Children's Hospital Institutional Review Board, (the committee that reviews all research involving human subjects at Nationwide Children's Hospital).



| Signature Block for Children | N/A, Adult Subject | |
|---|---|---|
| Your signature documents your permission for the named child t | o take part in this research. | |
| Printed name of child | _ | |
| Signature of parent or individual legally authorized to consent to the child's general medical care | <br>Date & Time | AM/PM |
| Printed name of parent or individual legally authorized to consento the child's general medical care | <del>T</del> | |
| Relationship to Participant | | |
| Note: Investigators are to ensure that individuals who are not particle consent to the child's general medical care. Contact Legal Servi | | al authority to |
| Signature of second parent or individual legally authorized to consent to the child's general medical care | Date & Time | AM/PM |
| Printed name of second parent or individual legally authorized to consent to the child's general medical care | _ | |
| Relationship to Participant | | |
| If signature of second parent not obtained, indicate why: (select □ Not required by IRB □ Second parent is deceased □ Second parent is unknown □ | | bly available |
| Signature of person obtaining consent | <br>Date & Time | AM/PM |
| Printed name of person obtaining consent | _ | |